CLINICAL TRIAL: NCT06440707
Title: Transcranial Electrical Stimulation in Stroke EaRly After Onset Clinical Trial 2
Brief Title: Transcranial Direct Current Stimulation for Treatment of Acute Ischemic Stroke
Acronym: TESSERACT 2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Johns Hopkins University (Other); Duke University (Other); Cedars-Sinai Medical Center (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mersedeh Bahr Hosseini, MD, Associate Professor of Neurology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-000780
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Cytoprotection; Collateral enhancement
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Adaptive Bayesian Design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Transcranial Direct Current Stimulation in patients ineligible for intravenous thrombolytic (Active Comparator): Patients in the active stimulation group receive cathodal transcranial electrical stimulation via 5 small electrodes for 20 to 60 minutes (min) at 1 or 2 milliamperes (mA) intensities. The duration and intensity of the stimulation will determined by the dose Tier the patient is assigned to. There will be 5 dose tiers, reflecting increasing intensity and duration of stimulation: Tier1- 2 mA, single 20 min cycle; Tier 2 - 1 mA, 2 cycles of 20 min/20 min off; Tier 3- 2mA, 2 cycles of 20 min/20 min off; Tier 4 - 1 mA, 3 cycles of 20min/20 min off; Tier 5 - 2 mA, 3 cycles of 20 min/20 min off.
  The decision to which dose Tier the patient should be assigned will be determined by the mathematical Bayesian model.
  Interventions: Device: High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS)
- Sham stimulation in patients ineligible for intravenous thrombolytic (Sham Comparator): Patients in the sham stimulation arm will have the cap and electrodes in place but will not receive electrical stimulation.
  Interventions: Device: Sham tDCS
- Transcranial Direct Current Stimulation in patients receiving intravenous thrombolytic (Active Comparator): Patients in the active stimulation group receive cathodal transcranial electrical stimulation via 5 small electrodes for 20 to 60 minutes (min) at 1 or 2 milliamperes (mA) intensities. The duration and intensity of the stimulation will determined by the dose Tier the patient is assigned to. There will be 5 dose tiers, reflecting increasing intensity and duration of stimulation: Tier1- 2 mA, single 20 min cycle; Tier 2 - 1 mA, 2 cycles of 20 min/20 min off; Tier 3- 2mA, 2 cycles of 20 min/20 min off; Tier 4 - 1 mA, 3 cycles of 20min/20 min off; Tier 5 - 2 mA, 3 cycles of 20 min/20 min off.
  The decision to which dose Tier the patient should be assigned will be determined by the mathematical Bayesian model.
  Interventions: Device: High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS)
- Sham stimulation in patients receiving intravenous thrombolytic (Sham Comparator): Patients in the sham stimulation arm will have the cap and electrodes in place but will not receive electrical stimulation.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: High-definition Cathodal Transcranial Direct Current Stimulation (HD C-tDCS) — The active study treatment involves delivering a weak form of electrical stimulation via 5 small electrodes to the brain tissue at risk of infarction.
  Arms: Transcranial Direct Current Stimulation in patients ineligible for intravenous thrombolytic; Transcranial Direct Current Stimulation in patients receiving intravenous thrombolytic
Device: Sham tDCS — Sham patients will have cap and electrodes in place, but no stimulation will be delivered.
  Arms: Sham stimulation in patients ineligible for intravenous thrombolytic; Sham stimulation in patients receiving intravenous thrombolytic

SUMMARY:
Many patients with acute ischemic stroke are ineligible for currently available standard treatments (clot-busting medication, also known as intravenous thrombolytic or mechanical removal of a clot), and many are non-responders, resulting in a low rate of excellent outcomes, which necessitates the development of novel therapies.

In this study, investigators are testing a new treatment in which a weak electrical current will be applied via scalp electrodes to increase collateral blood flow to the brain and rescue the brain tissue at risk of injury. The primary aim is to find an optimal dose of this therapy that is both adequately safe and effective on imaging markers of brain tissue rescue.

DETAILED DESCRIPTION:
This multi-site, phase 2a, randomized, sham-controlled, adaptive study aims to identify an optimal dose of a new treatment, cathodal direct current stimulation or C-tDCS, for acute ischemic stroke. This new treatment involves applying a weak inhibitory electrical current to the brain via scalp electrodes in acute stroke patients. The weak electrical current will electrically protect the brain cells not receiving enough oxygen and nutrients due to blood vessel blockage and increase the collateral blood flow to the brain.

The study primarily aims to find an optimal dose that shows adequate safety and effectiveness on markers of brain protection and collateral blood flow enhancement using brain scan. The investigators will ask acute stroke patients who arrive at the Emergency Departments of the University of California Los Angeles (UCLA), Duke, and Johns Hopkins Medical Center and are not candidates for clot removal procedure (endovascular thrombectomy) to participate in the study. The study enrolls patients in 2 subgroups depending on their eligibility for clot-busting medication, also known as thrombolytics (thrombolytic receiving and thrombolytic ineligible groups). Then, patients will be randomized in a 5 to 1 ratio to receive active stimulation versus sham (control with no stimulation).

Amongst patients randomized to the active arm, different doses of electrical current will be tested in various ranks, increasing the strength and the total duration of the electrical current at higher ranks. Computer simulation techniques (Bayesian method) will decide which dose patients should be assigned. The deciding rules of whether to escalate versus de-escalate versus stay on the same dose rank will be the probabilities of brain bleeding of ≤40% and substantial rescue of brain tissue at risk of permanent injury of ≥70%. The functional features and rules of the mathematical technique (Bayesian) will justify enrolling up to 50 patients in each subgroup of lytic-receiving and non-lytic-receiving patients (a total of up to 100 patients in active groups). Additionally, 10 sham (control) patients will be enrolled in each subgroup (a total of up to 20 patients in sham groups).

At 24-30 hours after the study stimulation, patients will receive a brain MRI to assess the presence of any brain bleed and how much brain tissue is rescued (primary aims), as well as to examine the additional effects of the study stimulation on brain collateral blood flow and the growth of the permanently damaged brain tissue.

As part of the study's additional goals, the treatment's tolerability will be studied by asking patients about how they feel during and after each session. Patients will also be neurologically examined after each session. Four days after enrollment, a brief neurological assessment will be performed if the patient is still in the hospital. On day 30, patients will receive a call from research personnel to see how they are doing. On day 90, they will be asked to come to neurology clinic to be neurologically assessed. The information gathered from this study will be used to advance this new treatment to future larger studies.

ELIGIBILITY:
Inclusion Criteria:

* New focal neurologic deficit consistent with AIS
* National Institute of Health Stroke Scale (NIHSS) ≥4 or NIHSS< 4 in the presence of disabling deficit (a deficit that, if unchanged, would prevent the
* patient from performing basic activities of daily living such as bathing, ambulating, toileting, hygiene, and eating or returning to work)
* Age>18
* Presence of any cortical vessel occlusion, including Internal Carotid Artery, branches of Middle Cerebral Artery, Anterior Cerebral Artery, Posterior Cerebral Artery, Posterior-Inferior Cerebellar Artery
* Presence of salvageable penumbra with perfusion lesion volume to ischemic core volume ratio of ≥ 1.2 on multimodal imaging
* Patient ineligible for endovascular thrombectomy per American Heart/Stroke Associations Guidelines
* Patient is able to be treated with tDCS within 24 hours of last known well time
* A signed informed consent is obtained from the patient or patient's legally authorized representative

Additional inclusion criteria for non-thrombolytic patients

• Patient ineligible for IV lytics per American Heart/American Stroke Associations National Guidelines

Additional inclusion criteria for thrombolytic receiving patients

* Patient eligible for tPA per Guidelines
* Within 2-hours from intravenous thrombolytic start of administration

Exclusion Criteria:

* Acute intracranial hemorrhage
* Presence of MRI and gadolinium contraindications including cardiac implantable devices, cochlear implant, implanted neurostimulation device, unremovable metallic body piercing, magnetic dental implants, drug infusion pumps, estimated glomerular filtration rate of less than 35 mL/min/1.73 m2, allergy to gadolinium
* Evidence of a large Ischemic core volume more than equal to 100 cc
* Presence of transcranial direct current stimulation contraindications - electrically or magnetically activated intracranial metal and non-metal implants.
* Pregnancy
* Signs or symptoms of acute myocardial infarction on admission
* History of seizure disorder or new seizures with presentation of current stroke
* Evidence of any other major life-threatening or serious medical condition that would prevent completion of the study protocol, including attendance at the 3-month follow-up visit
* Concomitant experimental therapy
* Preexisting scalp lesion at the site of the stimulation or presence of skull defects (may alter current flow
* pattern)
* Preexisting coagulopathy
* Patients suspected of having infective endocarditis and ischemic stroke related to septic emboli
* Patients suspected or known to be infected with coronavirus 2019 (COVID-19)
* Patient with radiographic evidence or suspicion of chronic conditions that may predispose them to intracranial hemorrhage, including brain arteriovenous malformations, cerebral cavernous malformations, cerebral telangiectasia, multiple previous intracerebral hemorrhages (amyloid angiopathy)
* Suspected cerebral vasculitis based on medical history and imaging
* Suspected cysticercosis
* Suspected cranial dural arteriovenous fistula
* Cerebral venous thrombosis
* Head trauma causing loss of consciousness, concussion, confusion, or a headache within the past 30 days
* Patient has suffered a hemorrhagic or ischemic stroke within the last three (3) months
* History of cancer known to cause hemorrhagic metastases, e.g., melanoma, renal cell carcinoma,
* choriocarcinoma, thyroid carcinoma, lung carcinoma, breast carcinoma, and hepatocellular carcinoma
* History of left atrial myxoma
* Evidence of dissection in the intracranial cerebral arteries
* Suspicion of aortic dissection
* Significant mass effect with midline shift
* The patient is in a coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Radiographic Intracranial Hemorrhage | At 24-30 hour post-stimulation
  Presence of any intracranial hemorrhage on brain MRI, including hemorrhagic infarction types 1,2 and parenchymal hematoma types 1 and 2.
Presence of Substantial Penumbra Salvage | At 24-30 hour post-stimulation
  Presence of substantial penumbra salvage on hemodynamic brain MRI is defined as the presence of salvage of more than equal to 40% of penumbra.

SECONDARY OUTCOMES:
Frequency of Symptomatic Intracranial Hemorrhage-Safety Outcome | At 24-30 hour post-stimulation
  Number of patients with parenchymal hemorrhage type 2 associated with worsening ≥ 4 on the National Institute of Health Stroke Scale (NIHSS)).
  The National Institute of Health Stroke Scale is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment; a higher score indicates worse neurological deficits.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (highest disability), with the minimum score being a 0 (lowest disability).
Frequency of Early Neurologic Deterioration-Safety Outcome | At 24-hour post-stimulation
  Number of patients with worsening of more than equal to 4 on the National Institute of Health Stroke Scale (NIHSS) during the 24-hour period after stimulation, with or without intracranial hemorrhage.
  The National Institute of Health Stroke Scale is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment; a higher score indicates worse neurological deficits.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (highest disability), with the minimum score being a 0 (lowest disability).
All-cause Mortality -Safety Outcome | At day 90 post-stimulation
  Number of patients with with outcome of death or modified Rankin Scale of 6
Frequency of Completion of Stimulation Protocol-Tolerability Outcome | At the end of each 20 minute stimulation period
  Number of participants who complete the protocol-assigned stimulation treatment without adverse effects as assessed by a modified Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events.
Frequency and Severity of Adverse Events-Tolerability Outcome | At the end of each 20 minute stimulation period
  Number of patients who experience adverse events as assessed by a modified Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events and severity of each event
Amount of Collateral Enhancement- Imaging Efficacy Biomarker Outcome | At 24-30 hour post-stimulation
  Percent change in the quantitative relative cerebral blood volume of the ischemic region as an index of collateral enhancement from baseline to post-stimulation
Infarct Core Growth- Imaging Efficacy Biomarker Outcome | At 24-30 hour post-stimulation
  Change in the infarct core volume in milliliters from baseline to post-stimulation
Reduction in Ischemic Lesion- Imaging Efficacy Biomarker Outcome | At 24-30 hour post-stimulation
  Change in perfusion lesion (ischemic lesion with Tmax>6sec) volume from baseline to post-stimulation

OTHER OUTCOMES:
Effect of Treatment on Rate of Intracranial Hemorrhage-Exploratory Efficacy Outcome | At 24-30 hour post-stimulation
  Number of active patients with intracranial hemorrhage on brain MRI, including hemorrhagic infarction types 1,2 and parenchymal hematoma types 1 and 2, compared to sham.
Effect of Treatment on Rate of Penumbral Salvage-Exploratory Efficacy Outcome | At 24-30 hour post-stimulation
  The amount of penumbra salvage, as assessed by hemodynamic brain MRI, in active patients will be compared to sham.
Early Neurological Improvement-Exploratory Early Clinical Efficacy Outcome | At 24-hour post-stimulation
  Number of patients with early neurological improvement as assessed by the National Institute of Health Stroke Scale.
  The National Institute of Health Stroke Scale is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment; a higher score indicates worse neurological deficits.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42 (highest disability), with the minimum score being a 0 (lowest disability).
Effect of Treatment on Disability- Exploratory Late Clinical Efficacy Outcome | At 90 days post-stimulation
  Improvement in disability is assessed by shift in the modified Rankin Scale.
  The modified Rankin Scale runs from 0-6, running from perfect health without symptoms (0) to death (6). A higher score indicates worse outcomes.
  0 - No symptoms.; 1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.
Dichotomized Assessment of Disability-Exploratory Late Clinical Efficacy Outcomes | At 90 days post-stimulation
  Number of patients with functional independence and non-disabled outcomes as assessed using the modified Rankin Scale.
  The modified Rankin Scale runs from 0-6, running from perfect health without symptoms (0) to death (6). A higher score indicates worse outcomes.
  0 - No symptoms.; 1 - No significant disability. Able to carry out all usual activities, despite some symptoms; 2 - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities; 3 - Moderate disability. Requires some help, but able to walk unassisted; 4 - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted; 5 - Severe disability. Requires constant nursing care and attention, bedridden, incontinent; 6 - Dead.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California- Los Angeles (UCLA), Los Angeles, California
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Duke Medical Center Hospital, Durham, North Carolina